CLINICAL TRIAL: NCT03821805
Title: Effects of Foot Reflexology Massage on Heart Rate Variability and Arterial Pulse Waveform After Yo Yo Intermittent Recovery Test and Repeated Sprint Test
Brief Title: Acute Effect of Foot Reflexology Massage on Heart Rate Variability and Arterial Pulse Waveform
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Taipei (Other)
Responsible Party: Principal Investigator, YUNG-SHENG CHEN, Associate Professor, University of Taipei
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UT-IRB-2016-017
Record Dates: First submitted 2019-01-22; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Massage; Anaerobic Exercise; Aerobic Exercise
Keywords: Heart rate variability; Arterial pulse waveform

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foot reflexology massage group (Experimental): The duration of intervention was 30 min (15 min massage duration for each leg)
  Interventions: Other: Foot reflexology massage
- Control group (No Intervention): Rest for 30 min

INTERVENTIONS:
Other: Foot reflexology massage — Foot reflexology technique of Father Josef was used as massage intervention
  Arms: Foot reflexology massage group

SUMMARY:
Foot reflexology treatment provides acute and chronic effects on cardiovascular and hemodynamic functions. However, no information is available to us in regarding the treatment effect of foot reflexology after exercise. This study investigated the acute effect of foot reflexology treatment on heart rate variability after anaerobic-based and aerobic-based intermittent exercises.

DETAILED DESCRIPTION:
The sympathetic activation and sympathy-vagal balance after repeat sprint performance can be immediately modulated by foot reflexology massage. The acute benefits of foot reflexology intervention on cardiac sympathovagal balance can be considered as exercise recovery strategies in sports.

ELIGIBILITY:
Inclusion Criteria:

* Undertake football/futsal training at least 3 times a week
* Age between 18 and 30 years old

Exclusion Criteria:

* History of severe neuromuscular injury
* Current lower extremity injury
* Current neurological diseases

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | immediately following intervention phase
  15 minutes resting electrocardiographic record at baseline and post-intervention phase

SECONDARY OUTCOMES:
Arterial pulse waveform | immediately following intervention phase
  15 minutes resting arterial plethysmographic waveform at baseline and post-intervention phase

IPD SHARING:
Plan to Share IPD: No
Individual participant data is protected by IRB application with a minimum of 3 years data storage.